CLINICAL TRIAL: NCT01357369
Title: Pharmacokinetics and Placental Transfer of Ondansetron and Cefazolin: A Preliminary Analysis
Brief Title: Study of Drug Concentration of Ondansetron and Cefazolin in Mothers and Neonates
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David R. Drover, Associate Professor, Stanford University
Other Study IDs: SU-02252011-7482; IRB 20231
Record Dates: First submitted 2011-05-10; First posted 2011-05-20 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Pregnancy Complications
Keywords: bacteria infections
MeSH Terms: conditions — Pregnancy Complications | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for pharmacokinetics.

GROUPS / COHORTS (1):
- Ondansetron/Cefazolin treatment: Pregnant women undergoing uncomplicated cesarean section deliveries who have consented to participate, and will receive Ondansetron and Cefazolin in the course of their clinical care will have PK blood samples drawn.
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Blood samples will be drawn from the mother, umbilical vein and artery post delivery, and neonate with other clinical labs.

SUMMARY:
This study proposes to look at the pharmacokinetics of two drugs (Cefazolin and ondansetron) given routinely to pregnant women who are planning to deliver via cesarean section. The investigators will evaluate the metabolism of both drugs by the pregnant woman, the placental transfer over time, and the subsequent metabolism of the transferred drug in the neonate.

DETAILED DESCRIPTION:
There is very little data on drug metabolism during pregnancy, and how it may differ from the non-pregnant woman. There is even less data on placental transfer of drug to the neonate when medications are given prior to delivery. This study proposes to look at the pharmacokinetics of two drugs (Cefazolin and ondansetron) given routinely to pregnant women who are planning to deliver via cesarean section. The investigators will evaluate the metabolism of both drugs by the pregnant woman, the placental transfer over time, and the subsequent metabolism of the transferred drug in the neonate.

The investigators hope to learn 1) the pk profile of both drugs in pregnancy, and how it differs from the non-pregnant woman, 2) the placental transfer of both drugs, and 3) the profile of neonatal metabolism of the drug that crosses the placental barrier.

ELIGIBILITY:
Inclusion Criteria:

Adult participant:

* Age 18-45 years old
* Term pregnancy (37-42 weeks)
* Delivers by planned cesarean section, or unplanned, non-urgent cesarean section.
* Generally healthy
* Able and willing to sign informed consent

Neonatal participant:

* Male of female
* 37-42 weeks gestation

Exclusion Criteria:

* Adult:Medical condition that would effect metabolism of the study drugs
* Known allergy to either study medication
* Use of medications in the last 48 hours that might induce or inhibit metabolism of ondansetron (e.g. barbiturates, fluconazole, erythromycin, etc.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Generally health women at 37-42 weeks gestation, and their newborns.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) results for Cefazolin and Ondansetron in maternal blood specimens | 10 hours
  Plasma concentrations will be reported in mg/L. Plasma concentration will then be analyzed using nonlinear mixed effects modeling (nonmem) software to determine volume of distribution in L and clearance in L/minute.

SECONDARY OUTCOMES:
Identification of placental transfer of studied meds (Cefazolin and Ondansetron) | 1 hr
  By measuring the PK of the studied drugs in the umbilical cord sample we hope to gain information regarding placental transfer.
  Plasma concentrations will be reported in mg/L. Plasma concentration will then be analyzed using nonlinear mixed effects modeling (nonmem) software to determine volume of distribution in L and clearance in L/minute.
PK results of neonatal blood specimens | 48 h
  Plasma concentrations will be reported in mg/L. Plasma concentration will then be analyzed using nonlinear mixed effects modeling (nonmem) software to determine volume of distribution in L and clearance in L/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, Sub-Investigator — Stanford University; David R. Drover, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States